CLINICAL TRIAL: NCT05338528
Title: Implementation and Assessment of the Elder-friendly BEdside Reconditioning for Functional ImprovemenTs (BE-FIT) Following Surgery Study
Brief Title: Implementation and Assessment of the BE-FIT Program
Acronym: BE-FIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00115917
Record Dates: First submitted 2022-04-10; First posted 2022-04-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Complications; Mobility; Surgery
Keywords: Exercise, Postoperative, Surgery
MeSH Terms: conditions — Postoperative Complications; Motor Activity

STUDY DESIGN:
Intervention Model Description: A quasi-experimental unblinded interrupted time-series (ITS) design in three phases: pre-intervention; during intervention; post-intervention. A before-and-after analysis methodology for complications, functional performance, and patient satisfaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BE-FIT (Experimental): The quasi-experimental unblinded interrupted time-series (ITS) design will be conducted in three phases: pre-intervention/ (10 weeks); during intervention (16 weeks); post-intervention (20 weeks). A cohort of patients on selected wards will receive the BE-FIT program intervention.
  Interventions: Behavioral: BE-FIT exercise program
- Usual care (No Intervention): We will adopt a before-and-after analysis methodology for complications, functional performance, and patient satisfaction. A control cohort of patients on the same ward will be compared to who received usual care prior to the intervention; this may include physiotherapy consultations ordered at the discretion of the surgical team or any other independent activity initiated by the patient (e.g., walking).

INTERVENTIONS:
Behavioral: BE-FIT exercise program — BE-FIT is an evidence-based exercise program that focuses on early mobilization and recovery by minimizing bed rest, promoting functional tasks, and encouraging self-management. The intervention ist based on the Mobilization of Vulnerable Elders (MOVE) program and consists of a bedside exercise plan, done independently by the patient without the need for additional rehabilitation or healthcare staff.
  Arms: BE-FIT

SUMMARY:
Lengthy hospitalization and immobility can lead to muscle loss resulting in reduced recovery rates and prolonged hospital stay or readmission. Older adults discharged from hospitals are at an increased risk for functional decline, falls and disability. Daily exercise and physical activities have proven to enhance the recovery and discharge process for older patients from the hospital and ultimately save vast amounts of dollars each year. The aim of this study is to initiate early mobilization and decrease the rate of functional decline in post-surgical older adults' patients in the acute care hospital setting in Alberta, Canada. The investigators are implementing a BE-FIT (BEdside reconditioning for Functional ImprovemenTs) a quality improvement, evidence-based exercise program that focuses on early mobilization and recovery by minimizing bed rest, promoting functional tasks, and encouraging self-management. Patients enrolled in the program will receive a bedside exercise plan to be completed independently throughout their stay in the hospital. Control patients will receive usual care without the added exercise plan. Patient mobility during their hospital stay will be assessed pre and post BE-FIT initiation according to a predetermined mobility scoring system. Secondary outcomes will include: time-to-mobility, length of stay, complication incidence and hospitalization costs.

DETAILED DESCRIPTION:
Frailty and post-operative complications are the predictors of increased cost-of-care among older patients who underwent emergency abdominal surgery in Alberta. In addition, older patients are often more vulnerable to the physical stressors following major surgery including risks of falls and disability. There is increasing evidence that daily exercise and physical activities can enhance the recovery and discharge process for older patients. Employing a two-arm trial design we will test whether the initiation of an early mobilization program can decrease the rate of functional decline in post-surgical older adults' patients.

The trial will be conducted in an acute care hospital setting in Alberta, Canada. The investigators will implement a quality improvement program BE-FIT (Bedside reconditioning for functional improvements) based on the Mobilization of Vulnerable Elders (MOVE) implementation strategy. BE-FIT is an evidence-based exercise program that focuses on early mobilization and recovery by minimizing bed rest, promoting functional tasks, and encouraging self-management. The intervention consists of a bedside exercise plan completed throughout the hospitalization. It is done independently without the need for additional rehabilitation or healthcare staff. The investigators will implement educational intervention to support the patients, staff, and families in bringing and sustaining change in practice and behavior from sedentary to physically active mobilization approach in the surgical area of the acute care setting. Control patients will receive usual care without the added exercise plan.

BE-FIT will be implemented in surgical units at 3 demonstrator sites (University of Alberta Hospital (UAH), Foothills Medical Centre (FMC) and the Misericordia Community Hospital (MCH)). Units may include General surgery, Otolaryngologic surgery, and Urology. The research will include all patients ≥65 years admitted to the hospital (emergency or elective) units.

The study is guided by the Knowledge-to-Action Cycle theory (K2A) and the Quality Implementation Framework (QIF) with interrupted time-series (IT) design. Prior to the implementation of the program, the investigators will used readiness assessments, identification of facilitators and barriers to post-operative mobility and co-designs with patients will be conducted. To measure and analyze the impact of our program, the primary outcome will evaluate the percentage of 'out of bed' occurrences as measured by an interrupted time series of mobility audits; secondary outcomes will include: time-to-mobility, length of stay, complication incidence and hospitalization costs. The quasi-experimental unblinded interrupted time-series (ITS) design will be conducted in three phases: pre-intervention (10 weeks); during intervention (16 weeks); post-intervention (20 weeks). A pre-intervention model will be created by using the first time-points over 10 weeks to analyze the primary outcome. To evaluate whether this model describes the baseline adequately, an estimate of the time-series models for the entire 84-time points (pre- and post-intervention) will be performed. To examine the impact of the BE-FIT exercise program on patient outcome, the investigators will use segmented linear regression models and correct the models for autocorrelation as required using the Cochrane-Orcutt method. This will be used to calculate the median daily length-of-stay for each week in the study period, classified into pre-, during and post-intervention. Regression methods will be used to assess mobilization outcome to investigate and compare the trend in median length-of-stay. A before-and-after analysis methodology will be adopted for complications, functional performance, and patient satisfaction. Regression models will be constructed using the parsimonious approach, multivariable linear (or transformed linear) regression, and logistic regression. Potential confounding baseline variables (i.e., age, sex, patient location before admission, admitting diagnosis, etc.) will be entered into the model and kept if deemed statistically (p<0.05) and/or clinically important. Health economic assessment will estimate mean cost for different sub-categories using appropriate regressions models for skewed cost data, adjusted for potential risk differences. The impact on patient's function and quality-of-life will be assessed with Short Performance Physical Battery (SPPB) and EQ-5D questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* age 65 or older
* patients admitted to hospital for surgical procedures such as general surgical, urologic, otolaryngologic, and transplant surgery

Exclusion Criteria:

* non-index admissions (i.e., transferred from another inpatient service)
* out-of-province
* palliative surgery
* multi-system trauma patients
* patients with a Clinical Frailty Scale score ≥ 7

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2180 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The change in percentage of 'Out of bed' observations | A quasi-experimental unblinded interrupted time-series (ITS) design will be conducted in three phases: pre-intervention/(10 weeks); during intervention (16 weeks); post-intervention (20 weeks).
  The primary outcome is the change in percentage of 'out of bed' observations among older surgery patients assessed for baseline audits (Pre-intervention), compared to audits in the intervention phase, and compared to audits post-intervention. The research team will perform visual audits 6 times/week (three times/day, two days/week or two times/day, three times/week), and will record patient identification numbers and types of mobility observed using the MOVE's audit tool. Frequencies (percentage) of out-of-bed will be compared to frequencies (percentage) of in-bed events.

SECONDARY OUTCOMES:
Time-to-mobility | within 20 weeks post intervention
  Time-to-mobility will be obtained from the patient charts. Shorter time-to-mobility indicates better health
Length of stay | within 20 weeks post intervention
  Length of stay will be obtained from the patient charts and DIMR. Reduced length of stay will indicate improved health
Complication incidence | within 20 weeks post intervention
  Complication incidence will be obtained as assessed by a post-operative morbidity survey and DIMR. Less complication incidence will indicate a beneficial outcome of the quality improvement initiative.
Hospitalization cost | within 20 weeks post intervention
  Hospitalization cost including in-hospital costs, readmissions at 30 days' post-discharge will be obtained by utilizing DIMR, Discharge Abstract Database and in-hospital micro-costing data from each site.
Patient satisfaction | within 20 weeks post intervention
  patient satisfaction will be assessed by a patient satisfaction questionnaire (PSQ-18)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel G Khadaroo, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD with other researchers outside the collaborator group

REFERENCES:
- [Background] Khadaroo RG, Warkentin LM, Wagg AS, Padwal RS, Clement F, Wang X, Buie WD, Holroyd-Leduc J. Clinical Effectiveness of the Elder-Friendly Approaches to the Surgical Environment Initiative in Emergency General Surgery. JAMA Surg. 2020 Apr 1;155(4):e196021. doi: 10.1001/jamasurg.2019.6021. Epub 2020 Apr 15. PMID 32049271
- [Background] Pederson JL, Padwal RS, Warkentin LM, Holroyd-Leduc JM, Wagg A, Khadaroo RG. The impact of delayed mobilization on post-discharge outcomes after emergency abdominal surgery: A prospective cohort study in older patients. PLoS One. 2020 Nov 6;15(11):e0241554. doi: 10.1371/journal.pone.0241554. eCollection 2020. PMID 33156849
- [Background] Hofmeister M, Khadaroo RG, Holroyd-Leduc J, Padwal R, Wagg A, Warkentin L, Clement F. Cost-effectiveness Analysis of the Elder-Friendly Approaches to the Surgical Environment (EASE) Intervention for Emergency Abdominal Surgical Care of Adults Aged 65 Years and Older. JAMA Netw Open. 2020 Apr 1;3(4):e202034. doi: 10.1001/jamanetworkopen.2020.2034. PMID 32242905
- [Background] McComb A, Warkentin LM, McNeely ML, Khadaroo RG. Development of a reconditioning program for elderly abdominal surgery patients: the Elder-friendly Approaches to the Surgical Environment-BEdside reconditioning for Functional ImprovemenTs (EASE-BE FIT) pilot study. World J Emerg Surg. 2018 May 21;13:21. doi: 10.1186/s13017-018-0180-7. eCollection 2018. PMID 29942346
- See also: Dr. Khadaroo's Reserach Website — http://sites.google.com/ualberta.ca/drkhadarooresearch/